CLINICAL TRIAL: NCT05107973
Title: The Effectiveness of Baduajin in People With Intellectual Disability in Supported Employment: A Randomized Clinical Controlled Trial
Brief Title: The Effectiveness of Baduajin in People With Intellectual Disability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, JON TORRES UNDA, Dr, Lecturer, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TORRES-UNDA 2021 BADUAJIN ID
Record Dates: First submitted 2021-07-25; First posted 2021-11-04 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Disability, Intellectual
Keywords: intellectual disability; sheltered work; ageing; function
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Intervention Model Description: Parallel Randomized Controlled Trail
Who Masked: Investigator
Masking Description: Randomization will be done by the person responsible for the project in the company. Nobody from the research team will know in which arm are enroled the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): in this arm of participants will be receiving the Baduajin intervention.
  Interventions: Other: Baduajin
- control (No Intervention): in this arm of participants will not receive any intervention

INTERVENTIONS:
Other: Baduajin — The intervention will consist in a 1 hour supervised Baduajin sessions conducted once a week a certified instructor with more than 10 years of experience. Each session will start with 5 min of warm up, 50 minutes of Baduajin and 5 min of cool down. In the main part the participants exercise the wholes set of Baduajin that consist of eigth forms.
  Arms: intervention

SUMMARY:
Due to the ageing process, individuals with intellectual disability (ID) experience decreased balance and loss of functionality at an earlier age than their peers without ID. Above-mentioned negative effects of the age affect particularly work ability, forcing to the retirement. It also implies difficulties for social interaction and economic problems, among others.

Baduajin is a traditional Chinese exercise and it has been demonstrated as an effective therapy in different alterations of the movement (i.e. Parkinson Disease).

The hypothesis of this study is that a training program of Badaujing will improve the balance and functionality of individuals with ID over 40 years old that from a company of in sheltered work.

Subjects with mild to moderate ID aged 40 years or older who are working in Lantegi Batuak (Bizkaia, Spain) will be invited to take part in an Baduajin intervention. The training program will consist in a 1 hour session each week during 9 month. Participants will be randomly assigned to a control or intervention group. Before and after the intervention, all the participants will be assessed with the following protocol: SPPB for functionality, balance in stabilometric platform, and strength of the upper limb.

DETAILED DESCRIPTION:
Intellectual disability (ID) is deﬁned as a signiﬁcantly reduced ability to understand new or complex information and to learn and apply new skills (impaired intelligence). This results in a reduced ability to cope independently (impaired social functioning), and begins before adulthood, with a lasting eﬀect on development. For the ﬁrst time in history, adults with intellectual and developmental disabilities are living to experience old age. Although the impact of ID on life expectancy is variable, most people with mild-to-moderate mental impairment can now expect to live as long as their non-disabled peers. Nevertheless, the ageing process and related functional problems seem to have an earlier onset in people with ID, charasterized by impairtment of movement and balance skills, which could lead to an increased risk of falls, and in turn, to a higher risk of disability and loss of quality of life.

The social and health-related beneﬁts of the integration of the people with ID in the workplace are well known. People with ID often want to participate in work and organisation. However, these persons are much less likely to be employed than their non-disabled peers. In addition, people with ID who are in employment tend to need to retire earlier, producing social, economic and health problems.

On one hand, Lantegi Batuak is a provider of supported employment for more than 1000 people with ID in Bizkaia (Spain). At the above-mentioend company it was found that workers with ID over 40 years old showed problems related to ageing, which include loss of body balance and in consequence less functionality. In consequence, methodologies for the prevention of the problems related to the ageing process in people with ID are particularlly interesting for the above-mentioned comapany, and can be potentially interesting for other public and private providers of supported employment. On the other hand, as has been previously demonstrated, Baduajing can enhance the body balance and functionality in different conditions. However, it have found no evidence concerning the use of this method for improving the function of people with ID.

The aim of this research is to ascertain the efficacy of a Baduanjing program for improving the body balance and functionality of people with ID, aged 40 or older, who are working in Lantegi Batuak. A total of 40 participants will be randomly allocated to a control or intervention group. The intervention will consist in a 1 hour supervised Baduajin group sessions conducted once a week during 9 month. The effect of the intervention and the lack of this will be assessed. For this, a full test-protocol including anthropometry, functionality and body balance, will be perform inmediatly before and after the intervention, as well as after 3 month of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Workers of Lantegi Batuak (Basque Country, Spain),
* Age: between 40 and 66 years old
* Diagnostic: mild to moderate ID or down syndrome, or Steinert disease
* Enough ability to participate in activities in groups of 10 people.

Exclusion Criteria:

* Previous experience in Baduajin
* Lack of capactiy to participate in groups.

Ages: 40 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Change of Functionality | Baseline (week 0), post-intervention (week 28) and 3 month after the intervention (week 40).
  Functionality assessed by the Short Physical Performance Battery.

SECONDARY OUTCOMES:
Change of Strength | Baseline (week 0), post-intervention (week 28) and 3 month after the intervention (week 40).
  Strength of the upper extremity assessed by the handgrip strength measured by a Jamar dynamometer
Change of Body Balance | Baseline (week 0), post-intervention (week 28) and 3 month after the intervention (week 40).
  Postural control is assessed with an stabilometric platform at an acquisition frequency of 50 Hz during 40 seconds.
Anthopometry | Baseline (week 0), post-intervention (week 28) and 3 month after the intervention (week 40).
  Height and body mass will be measured. Body Mass Index will be calculated as weight divided by height (kg/m2)

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Basque Country, Leioa, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Undecided